CLINICAL TRIAL: NCT01355562
Title: Phase II Trial of Outpatient Intravenous Interleukin-2 in Malignant Melanoma and Metastatic Kidney Cancer
Brief Title: Trial of Outpatient Intravenous Interleukin-2 in Malignant Melanoma and Metastatic Kidney Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary Investigator is no longer employed at LLU as of 02/29/12.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Chien-Shing Chen, M.D., Ph.D., Loma Linda University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5110062
Record Dates: First submitted 2011-04-28; First posted 2011-05-18 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Melanoma; Metastatic Kidney Cancer
MeSH Terms: conditions — Melanoma; Kidney Neoplasms | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interleukin-2 (IL-2) — Daily for 4 doses every 3 weeks for a total of 12 doses in an outpatient setting

SUMMARY:
The current study will test single agent IL-2 in stage IV melanoma and kidney cancer.

DETAILED DESCRIPTION:
The current study will test single agent IL-2 given daily for 4 doses every 3 weeks for a total of 12 doses in an outpatient setting in stage IV melanoma and kidney cancer to attempt to determine the response rate, how long the responses last, and median survival of this regimen in these two diseases. Responding patients and those with absence of disease progression may receive additional cycles of therapy every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic diagnosis of metastatic kidney cancer or malignant melanoma Patients may be either newly diagnosed with metastatic disease or may have received prior treatment for metastatic kidney cancer.
2. Patients must have measurable disease on physical exam or radiologic studies.
3. ECOG performance status of 0 or 1 and estimated survival of at least 3 months.
4. White blood count of > 3500/mm3, platelet count > 100,000/mm3, hemoglobin > 9.0 gm/dl; bilirubin, ALT, AST < 2 x upper limit of normal; serum creatinine < 2.0 mg/dl.
5. Patients must undergo a low-level cardiac stress test (or similar cardiac evaluation such as dobutamine stress echocardiogram or radionuclide-based stress test) for possible atherosclerotic heart disease. Patients with a positive stress test would be excluded from this trial.
6. Patients with elevated temperatures > 100.5 F must have sources of occult infection excluded.
7. Patients must be felt to have recovered from effects of prior therapy, such as > 2 weeks after prior chemotherapy.

Exclusion Criteria:

1. Medical illness requiring corticosteroids or other immunosuppressive agents (such as cyclosporin or methotrexate).
2. Autoimmune disease such as inflammatory arthritis, which could be exacerbated by immune-based therapy.
3. Prior history of psychiatric disorder, which could be exacerbated by interleukin-2.
4. Lactation or pregnancy.
5. Evidence of significant cardiovascular disease including history of recent (< 6 months prior) myocardial infarction, congestive heart failure, primary cardiac arrhythmias (not due to electrolyte disorder or drug toxicity, for example) beyond occasional PVC's, angina, positive low-level stress test, or cerebrovascular accident.
6. Current brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Response rate | 9 weeks

SECONDARY OUTCOMES:
how long the tumor shrinkage lasts | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter Quan, Jr., M.D., Principal Investigator — Loma Linda University Cancer Center
Locations (2):
- United States (2):
  - Highland Springs Medical Plaza, Beaumont, California
  - Loma Linda University Cancer Center, Loma Linda, California

REFERENCES:
- See also: Related Info — http://www.llucc.org